CLINICAL TRIAL: NCT05368987
Title: Neuromodulation of the Fear Extinction Circuit Using Temporally and Anatomically Specific TMS in Humans
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Mohammed Milad, Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HSC-MS-23-0426; R01MH125198 (NIH)
Record Dates: First submitted 2022-05-05; First posted 2022-05-10 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Fear Conditioning and Extinction Paradigm, plus Transcranial Magnetic Stimulation (TMS) (Experimental): Participants will undergo a 3-day experimental paradigm. On day 1, participants will undergo a resting-state and structural scans in the fMRI scanner. The data from this scan will be used to determine the specific location of the TMS target for each participant. And participants will be aversively conditioned to two cues in the fMRI scanner. Task based and resting-state scans will occur on this day.
  On day 2, subjects will undergo extinction training outside of the scanner where one of the conditioned cues will be paired with TMS in a temporally and anatomically specific manner. A resting-state scan will occur before and after inside the scanner.
  On day 3, conditioned cues will be presented during the extinction recall phase of the study. This phase will be conducted in the fMRI scanner. Task-based and resting-state scans will occur on this day.
  Interventions: Device: Transcranial magnetic stimulation (TMS); Behavioral: Fear Conditioning and Extinction Paradigm

INTERVENTIONS:
Device: Transcranial magnetic stimulation (TMS) — Research subjects will undergo non-invasive TMS, with a frequency of 20Hz and intensity of 120% of their resting motor threshold (rMT) at varying time points and locations.
Behavioral: Fear Conditioning and Extinction Paradigm — Participants will undergo a 3-day experimental paradigm. On day 1, participants will undergo a resting-state and structural scans in the fMRI scanner. The data from this scan will be used to determine the specific location of the TMS target for each participant. And participants will be aversively conditioned to two cues in the fMRI scanner. Task based and resting-state scans will occur on this day.
  On day 2, subjects will undergo extinction training outside of the scanner where one of the conditioned cues will be paired with TMS in a temporally and anatomically specific manner. A resting-state scan will occur before and after inside the scanner.
  On day 3, conditioned cues will be presented during the extinction recall phase of the study. This phase will be conducted in the fMRI scanner. Task-based and resting-state scans will occur on this day.

SUMMARY:
This study aims to explore the mechanisms of how transcranial magnetic stimulation (TMS) impacts fear circuits. The overarching objectives are to understand how varying TMS parameters affect targeted brain regions in order to optimize its impact on enhancing fear extinction memory consolidation in a population with known fear extinction deficiencies: post-traumatic stress disorder (PTSD). 250 subjects will take part in this research study across UTHealth Houston. The study will include preliminary screenings, baseline visits, and experimental visits across four days

DETAILED DESCRIPTION:
The experiments proposed are aimed to understand how timing and location of transcranial magnetic stimulation (TMS) in humans will impact their ability to reduce conditioned fear responses and impact the activation of their brain regions involved in fear regulation. The researchers will use a novel TMS approach to vary timing and location of its delivery so that the researchers can characterize and establish best time and location to obtain optimal impact on fear inhibition, and then test these parameters in PTSD patients and see if such can rescue extinction deficits in PTSD. The anticipated impact is to enhance our understanding of the neural mechanisms of associated with TMS use and explore potential novel approaches for advancing PTSD treatment.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent.
* Inclusion Criteria for PTSD Subjects - Diagnosis of current PTSD
* Inclusion Criteria: Healthy Controls (HC) - no current psychiatric disorders ("Axis I" disorders)

Exclusion Criteria:

* Lifetime history of seizure or significant head trauma or other significant neurologic disease (e.g., tic disorder)
* History of serious/significant psychiatric diagnoses ("Axis I" diagnoses)
* Current significant suicidal ideation, plan or intent or suicidal behavior in past 6 months based on CSSRS and clinical judgment or Self-injurious behavior that involves suicidal intent, requires medical attention, or occurs daily
* Use of neuroleptics within one year prior to study
* Current substance use
* Pregnancy (to be ruled out by urine β-HCG).
* Metallic implants or devices contraindicating magnetic resonance imaging.
* Currently taking medications that lower the seizure threshold. These include antipsychotics, high dose theophylline or stimulants such as methylphenidate. Patients taking bupropion must be on a stable dose (*last 3 months) and take less than or equal to 300 mg/day.
* Implanted devices in subject's head (shunts, cochlear implants); metal in subject's head (other than dental implants).
* High risk of adverse emotional or behavioral reaction, and/or an inability to understand study procedures or the informed consent process
* Additional exclusion criteria for Healthy controls (HC) group: Current psychiatric diagnosis ("Axis I" diagnosis)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Skin Conductance Response (SCR) | Experimental Day 1
  Conductance is measured by placing two electrodes next to the skin and passing a tiny electric charge between the two points. SCR is proportionally related to the number of sweat glands that are activated, meaning in essence that the more emotionally aroused an individual is, the more the SCR amount is increased.
Skin Conductance Response (SCR) | Experimental Day 3
  Conductance is measured by placing two electrodes next to the skin and passing a tiny electric charge between the two points. SCR is proportionally related to the number of sweat glands that are activated, meaning in essence that the more emotionally aroused an individual is, the more the SCR amount is increased.
Functional MRI (fMRI) blood-oxygen-level-dependent (BOLD) responses | Experimental Day 1
  fMRI data, including blood-oxygen-level-dependent (BOLD) responses, is used in neuroimaging studies assess neural correlate activations and observe the increase/decrease in activation of a particular brain area in response to a specific cue. When these cells are active, there is an increase in blood oxygen in the surrounding area.
Functional MRI (fMRI) blood-oxygen-level-dependent (BOLD) responses | Experimental Day 3
  fMRI data, including blood-oxygen-level-dependent (BOLD) responses, is used in neuroimaging studies assess neural correlate activations and observe the increase/decrease in activation of a particular brain area in response to a specific cue. When these cells are active, there is an increase in blood oxygen in the surrounding area.

SECONDARY OUTCOMES:
Score on State-Trait Anxiety Inventory (STAI) - Form Y1 | Experimental Day 1
  STAI - Form Y1 is a commonly used measure of trait and state anxiety that consists of 20 statements that describe oneself. Each statement is scored from 1 (Not at all) to 4 (very much so). The total score range is 20-80. STAI scores are commonly classified as "no or low anxiety" (20-37), "moderate anxiety" (38-44), and "high anxiety" (45-80).
Score on State-Trait Anxiety Inventory (STAI) - Form Y1 | Experimental Day 3
  STAI - Form Y1 is a commonly used measure of trait and state anxiety that consists of 20 statements that describe oneself. Each statement is scored from 1 (Not at all) to 4 (very much so). The total score range is 20-80. STAI scores are commonly classified as "no or low anxiety" (20-37), "moderate anxiety" (38-44), and "high anxiety" (45-80).

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Milad, PhD, Principal Investigator — The University of Texas Health Science Center at Houston (UTHealth Houston)
Locations (1):
- UTHealth Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data.Upon reasonable request. Requests should be directed to Mohammed.R.Milad@uth.tmc.edu. To gain access, data requestors will need to sign a data access agreement.